CLINICAL TRIAL: NCT03104647
Title: Evaluation of the Performance of VRP-Clinic in Healthy Subjects in the Support of Rehabilitation
Brief Title: VRP-Clinic Software Evaluation - in Support of Rehabilitation (VRP02)
Acronym: VRP02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VRHealth Group Ltd (Industry)
Collaborators: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VRP02-0076-17-SZMC
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VRP-Clinic (Experimental): VRP-Clinic software on a virtual reality platform
  Interventions: Other: VRP-Clinic

INTERVENTIONS:
Other: VRP-Clinic — Subjects will perform a series of neck movements guided by graphic instructions appearing in the virtual reality environment

SUMMARY:
The current study is designed to evaluate neck movements performed according to the VRP-Clinic software, and to verify that they promote physical activities that correspond with physical rehabilitation.

DETAILED DESCRIPTION:
The study will take place at Shaare Zedek Medical Center (SZMC). The study will include a single visit.

Each subject will put on the VR headset and perform a series of neck movements guided by graphic instructions appearing in the VR environment. The session will be recorded with a video camera which will subsequently be viewed and evaluated by clinicians. The clinicians will identify each movement seen on the video from a predefined list and determine if such a movement is recommended as part of a rehabilitation training program.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female
2. Age 18-65

Exclusion Criteria:

1. History of neck related disorders (Whiplash, disc degeneration disease or other acute cervical spine conditions)
2. Current neck pain
3. Under medical treatment or observation for any health-related issue during the study
4. Recent trauma
5. Oncology background
6. Acute disease/illness
7. Pregnancy.
8. Using drugs that could potentially affect physical function and balance (such as corticosteroids, antipsychotics or antidepressants)
9. Vision problems that require glasses (not all frame types can fit into the headset)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yair Barzilay, MD, Principal Investigator — Shaare Zedek Medical Center; Lilach Gavish, PhD, Study Director — Hebrew University of Jerusalem
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the Shaare ZedeK Medical Center during the 5th of July 2017.
Period: Overall Study
Arm/Group | VRP-Clinic
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VRP-Clinic
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of VRP-Clinic Neck Movements That the Assessing Clinician Recognizes as Rehabilitation Movements
Description: The movements are recorded on video and sent to clinicians for evaluation after the session is completed.
  The movements are then evaluated by the clinicians according to a predetermined list.
Time Frame: Up to 2 weeks after the session
Population: Each subject performed 8 movements and repeated them twice. Overall, 160 movements were performed by 20 subjects and repeated twice. The clinicians recognized all the movements and determined them as rehabilitation movements.
Measure: Number; unit: Movements
Units Other Than Participants: Movements
Arm/Group | VRP-Clinic
Number analyzed (Participants) | 20
Number analyzed (Movements) | 320
Movements | 320

2. Secondary Outcome: Number of Participants With Any Adverse Event Occurring During the Study
Description: Safety measure - The number of participants with any adverse event reported by the subject or observed by the investigator/clinician during the study will be recorded.
Time Frame: through study completion, an average of 2 weeks
Measure: Number; unit: participants
Arm/Group | VRP-Clinic
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: This was a single visit study with no follow up. The adverse event data was collected on the day of the visit.
Arm/Group | VRP-Clinic
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03104647/Prot_SAP_000.pdf